CLINICAL TRIAL: NCT04945681
Title: Evaluating the Effectiveness of a Pneumococcal Immunisation Campaign in a Camp for Internally Displaced People: A Non-randomised, Quasi-experimental Phase IV Intervention Study
Brief Title: Evaluating the Effectiveness of a Pneumococcal Immunisation Campaign in a Camp for Internally Displaced People
Acronym: EEPICC
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Save the Children (Other); Murdoch Childrens Research Institute (Other); Ministry of Health Development, Somaliland (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OPP1211787
Record Dates: First submitted 2021-06-14; First posted 2021-06-30 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Pneumococcal Infections
Keywords: Pneumococcal conjugate vaccine; Humanitarian; Crisis; Forced displacement; Mass vaccination; Quasi-experimental
MeSH Terms: conditions — Pneumococcal Infections | interventions — Pneumococcal Vaccines

STUDY DESIGN:
Intervention Model Description: Before vs. after quasi-experimental study. Entire study population of age-eligible children will be offered the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mass vaccination (Experimental): Mass vaccination of children aged 6 weeks to 4 years old with pneumococcal conjugate vaccine (PNEUMOSIL). Children 6 weeks to 11 months old receive two doses, spaced 4 weeks apart. All other children receive a single dose. Vaccination is simultaneous, as per a campaign delivery strategy.
  Interventions: Biological: Pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: Pneumococcal conjugate vaccine — Mass campaign offering simultaneous pneumococcal conjugate vaccination to all children aged below 5 years of age living in Digaale camp, Somaliland. Children aged below 12 months receive 2 doses of vaccine, spaced 4 weeks apart. All other children receive one dose.

SUMMARY:
Pneumococcal conjugate vaccine (PCV) is used routinely worldwide as part of infant immunisations to prevent acquisition of S. pneumoniae, the aetiologic agent responsible for a large proportion of early childhood pneumonia and invasive disease. However, PCV has seen minimal uptake in populations affected by forced displacement and humanitarian crises, where the burden of pneumococcal disease is plausibly elevated.

This study seeks to generate evidence on appropriate vaccination strategies for crisis-affected populations. The investigators plan to exhaustively vaccinate children aged between six months and four years in a camp for displaced persons outside Hargeisa, the capital of Somaliland. The study will deliver PCV in a campaign modality, so as to achieve both short- and long-term herd immunity effects that, the investigators hypothesise, will reduce population-wide nasopharyngeal S. pneumoniae transmission and thereby protect young children from pneumococcal disease.

The study will adopt a quasi-experimental design, with baseline and post-intervention surveys to evaluate changes in pneumococcal carriage, complemented by safety assessment in children aged over 2 years, who fall outside of the WHO prequalification age range for the vaccine that will be used in this study (i.e. PNEUMOSIL) and for whom PCV safety data are scarce. In addition, we the study will also collect longitudinal data on incidence of pneumonia and antibiotic prescriptions in the camp.

ELIGIBILITY:
Inclusion Criteria:

1. Resident in Digaale camp
2. Voluntary written/thumb-printed informed consent has been provided by a parent or caregiver
3. Subject's parent/caregiver must be able to comprehend and comply with study requirements and procedures
4. Subject's parents/caregivers must have a readily identifiable place of residence in the study area

Exclusion Criteria:

1. Known hypersensitivity to any component of any of the EPI vaccines, including diphtheria toxoid, in the child or any sibling
2. History of allergic disease or history of a serious reaction to any prior vaccination in the child or any sibling
3. History of anaphylactic shock, regardless of cause
4. History of long-term treatment (defined as 14 or more consecutive days) with immunosuppressants or other immune modifying drugs, including glucocorticoids, but excluding topical and inhaled glucocorticoids

Ages: 6 Weeks to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2882 (Actual)
Dates: Start 2022-11-27 (Actual); Primary Completion 2025-01-18 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Nasopharyngeal carriage of one or more colonies of vaccine-type Streptococcus pneumoniae serotypes in children below 24 months old | 6 months, relative to baseline (pre-vaccination)
  The outcome is determined at the individual level, through polymerase chain reaction (PCR) microarray analysis of nasal swab samples collected during a cross-sectional, population-representative sample survey of camp residents. The analysis will be stratified by age group (0-11 months, 12-23 months). Vaccine-type serotypes are defined as those that the Pneumosil vaccine (Serum Institute, India) is designed to provide immunity for, and include serotypes serotypes 1, 5, 6A, 6B, 7F, 9V, 14, 19A, 19F and 23F.
Nasopharyngeal carriage of one or more colonies of vaccine-type Streptococcus pneumoniae serotypes in children below 24 months old | 12 months, relative to baseline (pre-vaccination)
  The outcome is determined at the individual level, through PCR microarray analysis of nasal swab samples collected during a cross-sectional, population-representative sample survey of camp residents. The analysis will be stratified by age group (0-11 months, 12-23 months). Vaccine-type serotypes are defined as those that the Pneumosil vaccine (Serum Institute, India) is designed to provide immunity for, and include serotypes serotypes 1, 5, 6A, 6B, 7F, 9V, 14, 19A, 19F and 23F.
Nasopharyngeal carriage of one or more colonies of vaccine-type Streptococcus pneumoniae serotypes in children below 24 months old | 24 months, relative to baseline (pre-vaccination)
  The outcome is determined at the individual level, through PCR microarray analysis of nasal swab samples collected during a cross-sectional, population-representative sample survey of camp residents. The analysis will be stratified by age group (0-11 months, 12-23 months). Vaccine-type serotypes are defined as those that the Pneumosil vaccine (Serum Institute, India) is designed to provide immunity for, and include serotypes serotypes 1, 5, 6A, 6B, 7F, 9V, 14, 19A, 19F and 23F.
Number and proportion of vaccination recipients who experience solicited local and systemic adverse events following immunisation (AEFI) | within 7 days of receipt of each vaccine dose
  The outcome is determined at the individual level. 'Solicited' indicates that adverse events are identified by study staff using a pre-defined checklist of signs and symptoms and proactive monitoring or follow-up of vaccine recipients. AEFI will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) (version 24.0 or later). Outcome ascertainment will occur through (i) in-person monitoring of vaccine recipients for 30 minutes after vaccine administration, and (ii) exhaustive follow-up of all vaccine recipients 7 days after vaccination, with administration of a structured questionnaire to their parents or caregivers. All AEFI will be graded using a severity scale (0 - none; 1 - mild; 2 - moderate; 3- severe; 4 - very severe; 5 - fatal), and analysis will be stratified by severity and age group (6 weeks to 11 months old, 12 to 23 months old, 24 to 59 months old).
Number and proportion of vaccination recipients who experience solicited or unsolicited severe adverse events (SAE) following vaccination | within 7 days of receipt of each vaccine dose
  The outcome is determined at the individual level. SAE are defined as any AEFI with severity >= 3. Outcome ascertainment will occur through (i) in-person monitoring of vaccine recipients for 30 min after vaccine administration, (ii) exhaustive follow-up of all vaccine recipients 7 days after vaccination, with administration of a structured questionnaire to their parents or caregivers; (iii) availability of a 24/7 phone number which caregivers of vaccine recipients will be encouraged to contact; (iv) visits to the camp's single primary healthcare facility, during each day on which vaccination takes place, to identify any children presenting for care with a SAE; and (v) availability of a 24/7 phone number which clinicians at the primary healthcare facility will be encouraged to contact. Each SAE will be followed up until resolution. Relatedness of each SAE to vaccine receipt will be classified as 'unrelated', 'unlikely', 'possible', 'probable', 'definite' and 'not assessable'.

SECONDARY OUTCOMES:
Nasopharyngeal carriage of one or more colonies of vaccine-type Streptococcus pneumoniae serotypes in children and adults 24 months old or older | 6 months, relative to baseline (pre-vaccination)
  The outcome is determined at the individual level, through PCR microarray analysis of nasal swab samples collected during a cross-sectional, population-representative sample survey of camp residents. The analysis will be stratified by age group (24-59 months, 5 to 14 years, 15 to 29 years, 30 to 49 years, 50 years and above). Vaccine-type serotypes are defined as those that the Pneumosil vaccine (Serum Institute, India) is designed to provide immunity for, and include serotypes serotypes 1, 5, 6A, 6B, 7F, 9V, 14, 19A, 19F and 23F.
Nasopharyngeal carriage of one or more colonies of vaccine-type Streptococcus pneumoniae serotypes in children and adults 24 months old or older | 12 months, relative to baseline (pre-vaccination)
  The outcome is determined at the individual level, through PCR microarray analysis of nasal swab samples collected during a cross-sectional, population-representative sample survey of camp residents. The analysis will be stratified by age group (24-59 months, 5 to 14 years, 15 to 29 years, 30 to 49 years, 50 years and above). Vaccine-type serotypes are defined as those that the Pneumosil vaccine (Serum Institute, India) is designed to provide immunity for, and include serotypes serotypes 1, 5, 6A, 6B, 7F, 9V, 14, 19A, 19F and 23F.
Nasopharyngeal carriage of one or more colonies of vaccine-type Streptococcus pneumoniae serotypes in children and adults 24 months old or older | 24 months, relative to baseline (pre-vaccination)
  The outcome is determined at the individual level, through PCR microarray analysis of nasal swab samples collected during a cross-sectional, population-representative sample survey of camp residents. The analysis will be stratified by age group (24-59 months, 5 to 14 years, 15 to 29 years, 30 to 49 years, 50 years and above). Vaccine-type serotypes are defined as those that the Pneumosil vaccine (Serum Institute, India) is designed to provide immunity for, and include serotypes serotypes 1, 5, 6A, 6B, 7F, 9V, 14, 19A, 19F and 23F.
Nasopharyngeal carriage of one or more colonies of non-vaccine-type Streptococcus pneumoniae serotypes in children and adults | 6 months, relative to baseline (pre-vaccination)
  The outcome is determined at the individual level, through PCR microarray analysis of nasal swab samples collected during a cross-sectional, population-representative sample survey of camp residents. The analysis will be stratified by age group (0-11 months, 12-23 months, 24-59 months, 5 to 14 years, 15 to 29 years, 30 to 49 years, 50 years and above). Non-vaccine-type serotypes are defined as those that the Pneumosil vaccine (Serum Institute, India) is not designed to provide immunity for, i.e. any serotypes other than 1, 5, 6A, 6B, 7F, 9V, 14, 19A, 19F or 23F.
Nasopharyngeal carriage of one or more colonies of non-vaccine-type Streptococcus pneumoniae serotypes in children and adults | 12 months, relative to baseline (pre-vaccination)
  The outcome is determined at the individual level, through PCR microarray analysis of nasal swab samples collected during a cross-sectional, population-representative sample survey of camp residents. The analysis will be stratified by age group (0-11 months, 12-23 months, 24-59 months, 5 to 14 years, 15 to 29 years, 30 to 49 years, 50 years and above). Non-vaccine-type serotypes are defined as those that the Pneumosil vaccine (Serum Institute, India) is not designed to provide immunity for, i.e. any serotypes other than 1, 5, 6A, 6B, 7F, 9V, 14, 19A, 19F or 23F.
Nasopharyngeal carriage of one or more colonies of non-vaccine-type Streptococcus pneumoniae serotypes in children and adults | 24 months, relative to baseline (pre-vaccination)
  The outcome is determined at the individual level, through PCR microarray analysis of nasal swab samples collected during a cross-sectional, population-representative sample survey of camp residents. The analysis will be stratified by age group (0-11 months, 12-23 months, 24-59 months, 5 to 14 years, 15 to 29 years, 30 to 49 years, 50 years and above). Non-vaccine-type serotypes are defined as those that the Pneumosil vaccine (Serum Institute, India) is not designed to provide immunity for, i.e. any serotypes other than 1, 5, 6A, 6B, 7F, 9V, 14, 19A, 19F or 23F.
Mean bacteriological density of vaccine- and non-vaccine-type Streptococcus pneumoniae infections, among children and adults with at least one infecting colony in the nasopharynx | 6 months, relative to baseline (pre-vaccination)
  The outcome is determined at the individual level, through PCR microarray analysis of nasal swab samples collected during a cross-sectional, population-representative sample survey of camp residents. Bacteriological density is estimated after PCR analysis as copies per milliliter. The analysis will be stratified by age group (0-11 months, 12-23 months, 24-59 months, 5 to 14 years, 15 to 29 years, 30 to 49 years, 50 years and above), and by vaccine-type versus non-vaccine-type serotype colonies. Vaccine-type serotypes are defined as those that the Pneumosil vaccine (Serum Institute, India) is designed to provide immunity for, i.e. 1, 5, 6A, 6B, 7F, 9V, 14, 19A, 19F or 23F. Non-vaccine serotypes are defined as any other serotype.
Mean bacteriological density of vaccine- and non-vaccine-type Streptococcus pneumoniae infections, among children and adults with at least one infecting colony in the nasopharynx | 12 months, relative to baseline (pre-vaccination)
  The outcome is determined at the individual level, through PCR microarray analysis of nasal swab samples collected during a cross-sectional, population-representative sample survey of camp residents. Bacteriological density is estimated after PCR analysis as copies per milliliter. The analysis will be stratified by age group (0-11 months, 12-23 months, 24-59 months, 5 to 14 years, 15 to 29 years, 30 to 49 years, 50 years and above), and by vaccine-type versus non-vaccine-type serotype colonies. Vaccine-type serotypes are defined as those that the Pneumosil vaccine (Serum Institute, India) is designed to provide immunity for, i.e. 1, 5, 6A, 6B, 7F, 9V, 14, 19A, 19F or 23F. Non-vaccine serotypes are defined as any other serotype.
Mean bacteriological density of vaccine- and non-vaccine-type Streptococcus pneumoniae infections, among children and adults with at least one infecting colony in the nasopharynx | 24 months, relative to baseline (pre-vaccination)
  The outcome is determined at the individual level, through PCR microarray analysis of nasal swab samples collected during a cross-sectional, population-representative sample survey of camp residents. Bacteriological density is estimated after PCR analysis as copies per milliliter. The analysis will be stratified by age group (0-11 months, 12-23 months, 24-59 months, 5 to 14 years, 15 to 29 years, 30 to 49 years, 50 years and above), and by vaccine-type versus non-vaccine-type serotype colonies. Vaccine-type serotypes are defined as those that the Pneumosil vaccine (Serum Institute, India) is designed to provide immunity for, i.e. 1, 5, 6A, 6B, 7F, 9V, 14, 19A, 19F or 23F. Non-vaccine serotypes are defined as any other serotype.
Incidence rate of hospitalisations due to acute lower respiratory infection (ALRI) among children aged below 2 years of age | 24 months, relative to baseline (pre-vaccination)
  The outcome is determined at the population level, as a rate per person-time after division by the camp's estimated population of children aged below 2 years of age, updated through exhaustive census every 6 months. Hospitalisation is defined as admission of a child residing in the camp to a paediatric inpatient facility, with a final diagnosis of acute lower respiratory infection or pneumonia. The outcome is ascertained through a manual search of registers of all paediatric facilities that the camp population can realistically utilise, complemented by perusal of outpatient register records of the camp's single primary healthcare facility, to identify instances of children referred to hospitals. The diagnosis is as per clinical records. The outcome is ascertained retrospectively at baseline (vaccination campaign), and once every 6 months post-vaccination, for 24 months. However, only results after 24 months are analysed.
Rate of antibiotic prescription at outpatient care among children aged below 5 years of age | 24 months, relative to baseline (pre-vaccination)
  The outcome is determined at the aggregate (population) level, as a rate per person-time after division by the camp's estimated population of children aged below 5 years of age, which will also be updated through an exhaustive census every 6 months. The outcome is ascertained through consultation of the pharmacy register of the camp's single primary healthcare facility, by tallying the number of single prescriptions issued by the pharmacy to outpatients. Antibiotics are defined as per the World Health Organization's Model List of Essential Medicines. The outcome is ascertained retrospectively through record review conducted at baseline (vaccination campaign), and once every 6 months post-vaccination, for 24 months. However, only results after 24 months are analysed.
Proportion of the target population who receive the specified dosing regimen of pneumococcal conjugate vaccine during the vaccination campaign | Single time point - baseline (vaccination campaign)
  The outcome is determined at the individual level, but will be analysed at an aggregate (population) level, with stratification by age group (6 weeks to 11 months old, 12 to 23 months old, 24 to 59 months old, 5 to 14 years old). Before the vaccination campaign, all children aged 6 weeks old to 14 years old living in the camp will be systematically identified and registered. This list will serve as the denominator for the outcome, while the numerator will be children on the list who are successfully vaccinated, as per campaign administrative records. Successful vaccination is defined as injection with two doses of Pneumosil vaccine, spaced 4 weeks apart, in children aged 6 weeks to 11 months old, and one dose of Pneumosil vaccine in children aged 1 to 14 years old.

CONTACTS AND LOCATIONS:
Locations (1):
- Digaale internally displaced persons camp, Hargeisa, Hargeisa, Somaliland, Somalia

IPD SHARING:
Plan to Share IPD: Yes
Anonymised participant data will be deposited in a curated digital repository and made available subject to meeting access conditions.
Supporting Information: Analytic Code
Time Frame: June 2026 - May 2036
Access Criteria: Researchers wishing to apply for data should complete and submit a data application form, outlining the research purpose for which they wish to use the data, a list of variables that they wish to access, and information on how they fulfil the access conditions. If the application fulfils the eligibility criteria, the applicant will be provided with a Data Transfer Agreement that must be signed by their host organisation.
URL: https://datacompass.lshtm.ac.uk/information.html

REFERENCES:
- [Background] van Zandvoort K, Hassan AI, Bobe MO, Pell CL, Ahmed MS, Ortika BD, Ibrahim S, Abdi MI, Karim MA, Eggo RM, Ali SY, Hinds J, Soleman SM, Cummings R, McGowan CR, Mulholland EK, Hergeye MA, Satzke C, Checchi F, Flasche S. Pre-vaccination carriage prevalence of Streptococcus pneumoniae serotypes among internally displaced people in Somaliland: a cross-sectional study. Pneumonia (Nathan). 2024 Dec 5;16(1):25. doi: 10.1186/s41479-024-00148-6. PMID 39633426
- [Derived] McGowan CR, van Zandvoort K, Ibrahim SA, Hassan AI, Ahmed AM, Magan MA, Muhumed MH, Mohamed MS, Cummings R, Ali SY, Mohamed MA, Saed MA, Karim MA, Hergeye MA, Flasche S, Checchi F. Safety and coverage of Pneumosil pneumococcal polysaccharide conjugate vaccine (10-valent PCV) in a camp for internally displaced persons in Somaliland. Vaccine. 2026 Jan 1;69:127991. doi: 10.1016/j.vaccine.2025.127991. Epub 2025 Nov 19. PMID 41265006